CLINICAL TRIAL: NCT05599568
Title: Repeated Bout Effect i Neuromuscular Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mads Peter Godtfeldt Stemmerik (Other)
Responsible Party: Sponsor-Investigator, Mads Peter Godtfeldt Stemmerik, Subinvestigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P-2022-168
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Myopathy
MeSH Terms: conditions — Muscular Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise challenge (Other): At baseline, subjects will perform the selected exercise challenge followed by blood samples collected at rest and 0, 2, 4, 24 hours and 4 days after end of exercise. Muscle soreness will be measured by asking the participant how sore their muscles in their thighs are on a visual-analog scale (1-10) at the same timepoints. After 4 weeks (+/- 3 days) of normal daily activity, the same test will be performed including blood samples.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Either concentric or excentric exercise

SUMMARY:
The repeated bout effect (RBE) refers to the adaptation whereby a single bout of eccentric exercise protects against muscle damage from subsequent eccentric bouts. This effect has been shown in many muscle groups using both serum biomarkers, muscle soreness and imaging techniques. Though the effect is well described in healthy, it has never been studied in patients with neuromuscular diseases (NMDs).

In healthy, the RBE is only described using eccentric exercise, but unlike healthy persons, patients with NMDs can experience significant muscle damage with concentric exercise. This raises the question, if patients with NMDs could also show RBE when performing concentric exercise.

DETAILED DESCRIPTION:
The repeated bout effect (RBE) refers to the adaptation whereby a single bout of eccentric exercise protects against muscle damage from subsequent eccentric bouts. This effect has been shown in many muscle groups using both serum biomarkers, muscle soreness and imaging techniques. Though the effect is well described in healthy, it has never been studied in patients with neuromuscular diseases (NMDs).

NMDs are a common term for diseases that affect the muscles by disease processes in the motor neuron, peripheral nerve, neuromuscular junction or the muscles. The diseases can cause symptoms such as muscle weakness, muscle fatigue and sometimes muscle pain and varying degrees of physical disability. As the mechanisms for disease varies among NMDs, it is likely that some patients will experience RBE in a similar fashion to healthy, while others may not.

Recent years have shown significant breakthrough in the treatment development for various NMDs, and many of these treatments are currently or will soon be evaluated in clinical trials. As many trials will use exercise to evaluate treatment effect, it is vital to understand whether a single bout of exercise in itself provides a protective effect on the muscles of patients with NMDs.

In healthy, the RBE is only described using eccentric exercise, but unlike healthy persons, patients with NMDs can experience significant muscle damage with concentric exercise. This raises the question, if patients with NMDs could also show RBE when performing concentric exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* The ability to complete the exercise challenge
* No concurrent medical condition that could interfere with interpretation of the results
* Molecular diagnosis of the specific condition in specified patient groups or healthy control
* No active muscle injury on the test day (caused by recent exercise, seizures, trauma, etc.)

Exclusion Criteria:

* Cardiac or pulmonary disease contraindicating peak exercise testing or strenuous exercise defined as NYHA-class III-IV
* Veins that are too difficult to puncture for blood sampling, evaluated by the investigator
* Severe muscle weakness, that prevents the subject completing the exercise test, evaluated by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Delta CK | 1 month
  Change in peak kreatine kinase following first and second exercise bout.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromuscular Research Unit, 3342, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided